CLINICAL TRIAL: NCT02500550
Title: An Exploratory, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of a Two-dose Regimen of ATIR101, a T-lymphocyte Enriched Leukocyte Preparation Depleted ex Vivo of Host Alloreactive T-cells (Using Photodynamic Treatment), in Patients With a Hematologic Malignancy, Who Received a CD34-selected Hematopoietic Stem Cell Transplantation From a Haploidentical Donor
Brief Title: Safety and Efficacy of Two Doses of ATIR101, a T-lymphocyte Enriched Leukocyte Preparation Depleted of Host Alloreactive T-cells, in Patients With a Hematologic Malignancy Who Received a Hematopoietic Stem Cell Transplantation From a Haploidentical Donor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR-AIR-008
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: Haploidentical stem cell transplantation; Graft versus host disease; Immune reconstitution; Alloreactive T-cells; Photodynamic treatment; Hematologic malignancy; Transplant-related mortality
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATIR101 (Experimental)
  Interventions: Biological: ATIR101; Procedure: Haploidentical hematopoietic stem cell transplantation (HSCT); Procedure: TBI regime; Procedure: Non-TBI regime

INTERVENTIONS:
Biological: ATIR101 — T-lymphocyte enriched leukocyte preparation depleted ex vivo of host alloreactive T-cells (using photodynamic treatment). Two intravenous infusions with 2x10E6 viable T-cells/kg approximately 42 days apart (unless the second dose is reduced or halted for safety reasons).
Procedure: Haploidentical hematopoietic stem cell transplantation (HSCT) — CD34-selected HSCT from a haploidentical donor. In order to prepare the patient for the HSCT one of the following myeloablative conditioning regimens is recommended:
  * Total Body Irradiation (TBI) regime
  * Non-TBI regime
  (See below for details)
Procedure: TBI regime — * Fractionated TBI 200 cGy twice daily for 3 days on Day -10 to -8 (1200 cGy in 6 fractions)
  * Fludarabine 30 mg/m2 IV once daily for 5 days on Day -7 to -3
  * Thiotepa; 5 mg/kg IV twice daily for 1 day on Day -7
  * Anti-thymocyte globulin (ATG; Thymoglobulin®); 2.5 mg/kg once daily for 4 days on Day -5 to -2, as a continuous IV infusion for 8 hours. During the course of ATG, patients will receive methylprednisolone 2 mg/kg/day IV.
Procedure: Non-TBI regime — * Fludarabine; 30 mg/m2 IV once daily for 5 days on Day -8 to -4
  * Thiotepa; 5 mg/kg IV twice daily for 1 day on Day -7
  * Melphalan; 60 mg/m2 IV once daily for 2 days on Day -2 and -1
  * ATG (Thymoglobulin®); 2.5 mg/kg once daily for 4 days on Day -5 to -2, as a continuous IV infusion for 8 hours. During the course of ATG, patients will receive methylprednisolone 2 mg/kg/day IV.

SUMMARY:
The purpose of this study is to determine whether a repeat dose administration of ATIR101 is safe and effective when infused in patients with a hematologic malignancy following a T-cell depleted stem cell graft from a related haploidentical donor. All patients are planned to receive two ATIR101 doses of 2×10E6 viable T-cells/kg, unless the second dose is reduced or halted for safety reasons.

DETAILED DESCRIPTION:
Study CR-AIR-008 is an exploratory, open-label, multicenter study. After signing informed consent, patients will receive a hematopoietic stem cell transplantation (HSCT) from a related, haploidentical donor, followed by a first ATIR101 infusion at a dose of 2×10E6 viable T-cells/kg between 28 and 32 days after the HSCT. Patients will receive a second ATIR101 infusion at a dose of 2×10E6 viable T-cells/kg between 70 and 74 days after the HSCT. To evaluate safety of the second dose administration, the first 6 patients treated will be evaluated for the occurrence of dose limiting toxicity (DLT), defined as acute GvHD grade III/IV within 120 days post HSCT (or within 42 days after the second ATIR101 infusion in case of prior dose delays). If within the first 6 patients no DLT is observed, treatment of the remaining 9 patients will continue with two ATIR101 doses of 2×10E6 viable T cells/kg. If within the first 6 patients at least 2 patients show DLT, the second ATIR101 infusion will be adjusted to a dose of 1×10E6 viable T cells/kg. If in one of the next 3 patients treated at this lower dose again DLT is observed, the second ATIR101 infusion will be halted and the remaining patients will be given only a single dose of ATIR101.

All patients treated with ATIR101 will be followed up until 12 months after the HSCT. Assessments will be performed at weekly visits from the day of the first ATIR101 infusion (Week 4) until 6 weeks after the second ATIR101 infusion (Week 16), at monthly visits from 4 until 6 months after the HSCT, and every 3 months from 6 until 12 months after the HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following hematologic malignancies:

  * Acute myeloid leukemia (AML) in first remission with high-risk features or in second or higher remission
  * Acute lymphoblastic leukemia (ALL) in first remission with high-risk features or in second or higher remission
  * Myelodysplastic syndrome (MDS): transfusion-dependent, or intermediate or higher IPSS-R risk group
* Karnofsky performance status ≥ 70%
* Eligible for haploidentical stem cell transplantation according to the investigator
* Male or female, age ≥ 18 years and ≤ 65 years

Exclusion Criteria:

* Availability of a fully matched related or unrelated donor following a donor search
* Diffusing capacity for carbon monoxide (DLCO) < 50% predicted
* Left ventricular ejection fraction < 50% (evaluated by echocardiogram or MUGA)
* AST > 2.5 x ULN (CTCAE grade 2)
* Bilirubin > 1.5 x ULN (CTCAE grade 2)
* Creatinine clearance < 50 mL/min (calculated or measured)
* Positive HIV test
* Positive pregnancy test (women of childbearing age only)
* Prior allogeneic HSCT
* Estimated probability of surviving less than 3 months
* Known allergy to any of the components of ATIR101 (e.g., dimethyl sulfoxide)
* Known presence of HLA antibodies against the non-shared donor haplotype
* Any other condition which, in the opinion of the investigator, makes the patient ineligible for the study

Inclusion Criteria Donor:

* Haploidentical family donor with 2 to 3 mismatches at the HLA-A, -B and/or -DR loci of the unshared haplotype
* Male or female, age ≥ 16 and ≤ 75 years (If applicable, local legal requirements for donors under the age of 18 will be followed)
* Eligible for donations of human blood and blood components according to local requirements and regulations
* Eligible for donation according to the transplantation center

Exclusion Criteria Donor:

* Positive pregnancy test or nursing (women of childbearing age only)
* Positive viral test for HIV-1, HIV-2, HBV, HCV, Treponema pallidum, HTLV 1 (if tested), HTLV-2 (if tested), or WNV (if tested)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Claude Roy, Prof MD, Principal Investigator — Maisonneuve-Rosemont Hospital (Montreal, Canada); Stephan Mielke, Prof MD, Principal Investigator — Centre for Allogeneic Stem Cell Transplantation, Karolinska University Hospital (Stockholm, Sweden)
Locations (11):
- Belgium (4):
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Canada (2):
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- University Hospital Centre Zagreb, Zagreb, Croatia
- University Medical Center Mainz, Mainz, Germany
- Hospital de Santa Maria, Clinica Universitaria Hematologia, Lisbon, Portugal
- United Kingdom (2):
  - Heartlands Hospital, Birmingham
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ATIR101: ATIR101: T-lymphocyte enriched leukocyte preparation depleted ex vivo of host alloreactive T-cells (using photodynamic treatment). Two intravenous infusions with 2x10E6 viable T-cells/kg approximately 42 days apart (unless the second dose is reduced or halted for safety reasons).
  Haploidentical hematopoietic stem cell transplantation (HSCT): CD34-selected HSCT from a haploidentical donor. In order to prepare the patient for the HSCT one of the following myeloablative conditioning regimens is recommended:
  * Total Body Irradiation (TBI) regime
  * Non-TBI regime
  (See below for details)
  TBI regime: • Fractionated TBI 200 cGy twice daily for 3 days on Day -10 to -8 (1200 cGy in 6 fractions)
  * Fludarabine 30 mg/m2 IV once daily for 5 days on Day -7 to -3
  * Thiotepa; 5 mg/kg IV twice daily for 1 day on Day -7
  * Anti-thymocyte globulin (ATG; Thymoglobulin®); 2.5 mg/kg once daily for 4 days on Day -5 to -2, as a continuous IV infusion for 8 hours. During the course of ATG, patients will receive methylprednisolone 2 mg/kg/day IV.
  Non-TBI regime: • Fludarabine; 30 mg/m2 IV once daily for 5 days on Day -8 to -4
  * Thiotepa; 5 mg/kg IV twice daily for 1 day on Day -7
  * Melphalan; 60 mg/m2 IV once daily for 2 days on Day -2 and -1
  * ATG (Thymoglobulin®); 2.5 mg/kg once daily for 4 days on Day -5 to -2, as a continuous IV infusion for 8 hours. During the course of ATG, patients will receive methylprednisolone 2 mg/kg/day IV.
Period: Overall Study
Arm/Group | ATIR101
Started | 15
Completed | 8
Not Completed | 7
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Arm/Group | ATIR101
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 41 [15 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7
  Belgium | 5
  United Kingdom | 2
  Germany | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Graft Versus Host Disease (GVHD) Grade III/IV
Time Frame: 180 days post HSCT
Population: The primary study endpoint, grade III/IV acute GVHD within 180 days after HSCT, was met for two patients treated with two doses of ATIR101.
  Two patients developed grade III/IV acute GVHD within 180 days after HSCT treated with a single dose of ATIR101.
Measure: Number; unit: participants
Arm/Group | ATIR101
Number analyzed (Participants) | 15
participants
  Single dose of ATIR101, grade III/IV acute GVHD within 180 days after HSCT: number analyzed (Participants) | 9
  Single dose of ATIR101, grade III/IV acute GVHD within 180 days after HSCT | 2
  Two doses of ATIR101, Grade III/IV acute GVHD within 180 days after HSCT: number analyzed (Participants) | 6
  Two doses of ATIR101, Grade III/IV acute GVHD within 180 days after HSCT | 2

2. Secondary Outcome: Incidence and Severity of Acute and Chronic GVHD
Time Frame: Between 6 and 12 months after HSCT
Population: 7 patients in the single dose and 4 patients in the double dose were analysed to make a total of 11 patients analysed.
Measure: Number; unit: Participants
Arm/Group | ATIR101
Number analyzed (Participants) | 11
Participants
  Single dose group acute GVHD between 6 and 12 months after HSCT: number analyzed (Participants) | 7
  Single dose group acute GVHD between 6 and 12 months after HSCT | 0
  Double dose group acute GVHD between 6 and 12 months after HSCT: number analyzed (Participants) | 4
  Double dose group acute GVHD between 6 and 12 months after HSCT | 0
  Single dose group chronic GVHD between 6 and 12 months after HSCT: number analyzed (Participants) | 7
  Single dose group chronic GVHD between 6 and 12 months after HSCT | 0
  Double dose group chronic GVHD between 6 and 12 months after HSCT: number analyzed (Participants) | 4
  Double dose group chronic GVHD between 6 and 12 months after HSCT | 2

3. Secondary Outcome: Percentage of Participants Who Achieved T-Cell Reconstitution at 6 and 12 Months Post HSCT
Description: Defined as CD3+ in peripheral blood higher than 0.2×10E9/L at 6 and 12 months post HSCT.
Time Frame: 6 and 12 months post HSCT
Population: Cumulative incidence estimates of T-cell reconstitution at 6 and 12 months post HSCT were analyzed for the single dose group (N=9) and double dose group (N=6).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATIR101
Number analyzed (Participants) | 15
percentage of participants
  Cumulative incidence estimates of T-cell reconstitution, 6 months post HSCT. Single dose group.: number analyzed (Participants) | 9
  Cumulative incidence estimates of T-cell reconstitution, 6 months post HSCT. Single dose group. | 44.4 [11.0 to 74.2]
  Cumulative incidence estimates of T-cell reconstitution, 6 months post HSCT. Double dose group.: number analyzed (Participants) | 6
  Cumulative incidence estimates of T-cell reconstitution, 6 months post HSCT. Double dose group. | 50.0 [8.2 to 82.6]
  Cumulative incidence estimates of T-cell reconstitution, 12 months post HSCT. Single dose group.: number analyzed (Participants) | 9
  Cumulative incidence estimates of T-cell reconstitution, 12 months post HSCT. Single dose group. | 77.8 [32.7 to 94.5]
  Cumulative incidence estimates of T-cell reconstitution, 12 months post HSCT. Double dose group.: number analyzed (Participants) | 6
  Cumulative incidence estimates of T-cell reconstitution, 12 months post HSCT. Double dose group. | 50.0 [8.2 to 82.6]

4. Secondary Outcome: Viral, Fungal, and Bacterial Infections
Description: Infection was defined as (1) a clinically apparent infectious disease with symptoms or (2) a viral reactivation. Severity was graded according to CTCAE vs. 4.0
Time Frame: From 6 months to 1 year after HSCT
Measure: Number; unit: Participants
Arm/Group | ATIR101
Number analyzed (Participants) | 11
Participants
  Any infection | 10
  Severity, grade 1-2 | 7
  Severity, grade 3-5 | 3

5. Secondary Outcome: Transplant-related Mortality (TRM)
Description: Defined as death due to causes other than disease relapse or progression, or other causes which are unrelated to the transplantation procedure (e.g. accident, suicide)
Time Frame: 12 months post HSCT
Population: Nine participants received a single dose of ATIR101 and 6 participants received a double dose of ATIR101
Measure: Number (95% Confidence Interval); unit: percentage of participants that died
Arm/Group | ATIR101
Number analyzed (Participants) | 15
percentage of participants that died
  Single-dose group, cumulative estimates of TRM: number analyzed (Participants) | 9
  Single-dose group, cumulative estimates of TRM | 22.2 [2.8 to 53.3]
  Double-dose group, cumulative estimates of TRM: number analyzed (Participants) | 6
  Double-dose group, cumulative estimates of TRM | 66.7 [12.2 to 92.5]

6. Secondary Outcome: Relapse-related Mortality (RRM)
Description: Defined as death due to disease relapse or disease progression
Time Frame: 12 months post HSCT
Population: Nine participants received a single dose of ATIR101 and 6 participants received a double dose of ATIR101
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATIR101
Number analyzed (Participants) | 15
percentage of participants
  Single dose group, cumulative estimates of RRM 12 months post HSCT: number analyzed (Participants) | 9
  Single dose group, cumulative estimates of RRM 12 months post HSCT | 11.1 [0.5 to 40.9]
  Double dose group, cumulative estimates of RRM 12 months post HSCT: number analyzed (Participants) | 6
  Double dose group, cumulative estimates of RRM 12 months post HSCT | 0 [0 to 0]

7. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from HSCT until death from any cause
Time Frame: 12 months post HSCT
Population: Nine participants received a single dose of ATIR101 and 6 participants received a double dose of ATIR101
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ATIR101
Number analyzed (Participants) | 15
Percentage of participants
  Single dose group, Kaplan-Meier estimates of OS 12 months post HSCT: number analyzed (Participants) | 9
  Single dose group, Kaplan-Meier estimates of OS 12 months post HSCT | 66.7 [28.2 to 87.8]
  Double dose group, Kaplan-Meier estimates of OS 12 months post HSCT: number analyzed (Participants) | 6
  Double dose group, Kaplan-Meier estimates of OS 12 months post HSCT | 33.3 [4.6 to 67.6]

8. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from HSCT until relapse, disease progression, or death, whichever occurs first
Time Frame: 12 months post HSCT
Population: Nine participants received a single dose of ATIR101 and 6 participants received a double dose of ATIR101
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ATIR101
Number analyzed (Participants) | 15
Percentage of participants
  Single dose group, Kaplan-Meier estimates of PFS 12 months post HSCT: number analyzed (Participants) | 9
  Single dose group, Kaplan-Meier estimates of PFS 12 months post HSCT | 55.6 [20.4 to 80.5]
  Double dose group, Kaplan-Meier estimates of PFS 12 months post HSCT: number analyzed (Participants) | 6
  Double dose group, Kaplan-Meier estimates of PFS 12 months post HSCT | 33.3 [4.6 to 67.6]

9. Secondary Outcome: GVHD-free, Relapse-free Survival (GRFS)
Description: Defined as the time until acute GVHD grade III/IV, chronic GVHD requiring systemic treatment, relapse, or death, whichever occurs first
Time Frame: 12 months post HSCT
Population: Nine subjects received a single dose of ATIR101 and 6 subjects received a double dose of ATIR101.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ATIR101
Number analyzed (Participants) | 15
Percentage of participants
  Single dose, Kaplan-Meier estimates of GRFS: number analyzed (Participants) | 9
  Single dose, Kaplan-Meier estimates of GRFS | 55.6 [20.4 to 80.5]
  Double dose, Kaplan-Meier estimates of GRFS: number analyzed (Participants) | 6
  Double dose, Kaplan-Meier estimates of GRFS | 16.7 [0.8 to 51.7]

ADVERSE EVENTS:
Time Frame: The median follow-up time of ATIR101-treated patients in the study was 11.6 (range 2.7-12.8) months after hematopoietic stem cell transplantation (HSCT) .
Arm/Group | ATIR101
All-Cause Mortality (participants affected / at risk) | 7/15
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATIR101 (N=15)
Acute graft-versus-host disease (GVHD) (Immune system disorders) | 5
Chronic GVHD (Immune system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATIR101 (N=15)
Acute GVHD (Immune system disorders) | 7
Chronic GVHD (Immune system disorders) | 2
Cytomegalovirus (CMV) positive (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02500550/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT02500550/SAP_001.pdf